CLINICAL TRIAL: NCT00061347
Title: Trans-Rectal Placement of Prostatic Fiducial Markers Under MR-Guidance in Patients Receiving External Beam Radiotherapy for Prostate Cancer: A Pilot Study
Brief Title: Using Fiducial Markers to Aid in Prostate Cancer Radiation Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 030190; 03-C-0190; NCT00882349 (obsolete NCT alias)
Record Dates: First submitted 2003-05-23; First posted 2003-05-26 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04-19

CONDITIONS: Prostate Cancer; Cancer
Keywords: Fiducial Marker; MRI; Prostate Cancer; Radiation
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

ARMS (1):
- 1 (Experimental): Placement of fidicual markers under MRI guidance for localization of radiaiton treatment
  Interventions: Procedure: Fiducial marker placement

INTERVENTIONS:
Procedure: Fiducial marker placement — Placement of fidicual markers under MRI guidance for localization of radiaiton treatment

SUMMARY:
To effectively treat prostate cancer, doctors need an accurate view (via X-rays) of the prostate gland during radiation therapy. To help improve this view, doctors may insert gold markers called fiducials into the prostate by placing hollow gold needles through the rectum and moving a fiducial through each needle. The purpose of the study is to determine whether an MRI scan can help doctors improve their placement of these needles.

Fifteen men will participate in this study. Patients will take the antibiotic levofloxacin for two days prior to the placement of the fiducials, then will have a small enema and another dose of the antibiotic on the morning of the procedure. After being anesthetized, patients will have an antenna-like tube placed into the rectum and have MRI images taken of the area. The doctor will then use these scans to place four fiducials into the prostate. The procedure will require approximately 45 minutes. Patients will be allowed to go home the same day of the procedure, which will be followed by a seven-week course of standard radiation therapy.

Prior to their participation in this study, patients will undergo the following evaluations: a physical exam, blood work, urine tests, and, if appropriate, an MRI or bone scan.

DETAILED DESCRIPTION:
Effective image-guided prostate therapies require excellent visualization of the prostate and surrounding anatomy, such that cancerous tissue can be treated while avoiding nearby neural and vascular structures. As such, Magnetic Resonance Imaging is well suited for image-guidance because of its excellent soft tissue contrast, multiplanar capabilities, and the potential to yield spectral/biological tumor mapping. Despite the potential for MRI-guided prostate therapies, there are currently no techniques that allow for precise trans-rectal intraprostatic needle placement in patients.

In this pilot study we seek to validate the accuracy and tolerability of a new system and technique that allows for accurate placement of needles within the prostate based upon MR images. The method is very similar to transrectal ultrasound guided biopsy of the prostate, except that it is applicable within a closed high-field MRI scanner. Four gold fiducial markers will be placed within the prostate under needle guidance in a series of patients with localized prostate cancer before external beam radiotherapy. Fifteen patients will be enrolled onto this study with sample size determined to obtain reasonably precise estimates of mean placement accuracy. The accrual period is expected to be less than a year.

While placement of the fiducial markers has no direct therapeutic benefit for the patient, intraprostatic radiopaque fiducial markers (placed under ultrasound) have shown value in assessing daily setup errors and off-line organ motion during external beam radiation therapy for prostate cancer. Therefore, a secondary objective is to gain experience using these intraprostatic fiducial markers for daily assessment and adjustment of external radiation beam targeting. These markers can also be utilized to aid in CT-MRI fusion and results in better target delineation for treatment planning. In this way, prostate cancer patients who are receiving external-beam radiation therapy may benefit from participation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Pathologically confirmed adenocarcinoma of the prostate gland.
* Age greater than or equal to 18 years.
* ECOG performance status of 0 or 1.
* Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed (this does not include routine laboratory tests or imaging studies required to establish eligibility).

EXCLUSION CRITERIA:

Patients with contraindication to transrectal needle placement:

* Bleeding disorder;
* PT/PTT greater than 1.5.times the upper limit of normal;
* Platelets less than 50K;
* Artificial heart valve.

Patients with contraindications to MRI:

* Patients weighing greater than 136 kg (weight limit for scanner table);
* Patients with pacemakers, cerebral aneurysm clips, shrapnel injury, or implanted electronic devices.
* Patients with chronic inflammatory bowel disease.
* Patients with distant metastatic disease.
* Patients with a prior history of pelvic or prostate radiotherapy.
* Cognitively impaired patients who cannot give informed consent.
* Other medical conditions deemed by the PI or associates to make the patient ineligible for protocol investigations, procedures, and high-dose external beam radiotherapy.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-05-23; Primary Completion 2004-05-31 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that MRI guidance allows for accurate fiducial marker placement within the prostate | 1, 3, 6, 12, 18, 24, 36, 48, and 60 months
To determine the toxicity of MR-Guided fiducial marker placement | 1, 3, 6, 12, 18, 24, 36, 48, and 60 months

SECONDARY OUTCOMES:
To gain preliminary experience using intraprostatic fiducial markers for daily set-up assessment and adjustment of external radiation beam targeting. | completion of study
To gain preliminary experience using intraprostatic fiducial markers for image fusion. | completion of study
To measure the magnitude of marker migration during the course of radiotherapy. | completion of study
To gather data on radiation therapy effects on prostate cancer patients treated at the NCI ROB. | completion of study
To gather data on the feasibility, tolerability, and effectiveness of local anesthetic injection along the neurovascular bundle under MRI guidance. | completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Yu KK, Hricak H. Imaging prostate cancer. Radiol Clin North Am. 2000 Jan;38(1):59-85, viii. doi: 10.1016/s0033-8389(05)70150-0. PMID 10664667
- [Background] Knopp MV, Weiss E, Sinn HP, Mattern J, Junkermann H, Radeleff J, Magener A, Brix G, Delorme S, Zuna I, van Kaick G. Pathophysiologic basis of contrast enhancement in breast tumors. J Magn Reson Imaging. 1999 Sep;10(3):260-6. doi: 10.1002/(sici)1522-2586(199909)10:33.0.co;2-7. PMID 10508285
- [Background] Kurhanewicz J, Vigneron DB, Hricak H, Narayan P, Carroll P, Nelson SJ. Three-dimensional H-1 MR spectroscopic imaging of the in situ human prostate with high (0.24-0.7-cm3) spatial resolution. Radiology. 1996 Mar;198(3):795-805. doi: 10.1148/radiology.198.3.8628874.